CLINICAL TRIAL: NCT00611728
Title: A Phase I Study of SU011248 Plus Irinotecan in the Treatment of Patients With Malignant Glioma
Brief Title: Ph I SU011248 + Irinotecan in Treatment of Pts w MG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000931
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2011-12

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; CPT 11; Sutent; Sunitinib; Sunitinib malate; Malignant Glioma; GBM; Irinotecan; Camptosar; Anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligoastrocytoma; SU011248; Brain tumor; Recurrent malignant glioma
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Oligodendroglioma; Brain Neoplasms | interventions — Sunitinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SU011248 & Irinotecan — Sutent given in daily oral manner for 1st 4 wks of each 6wk cycle. You will not take any Sutent during last 14 days of each 6 wk cycle. CPT-11 will be given intravenously over 1 & 1/2 hrs on 1st day of each cycle & then again on days 14 & 28.
  Sutent is approved for adult subjects w some forms of kidney cancer. It is considered "investigational" for brain tumors. Dosing will begin on day 1 of cycle 1 & continue daily for 4 wks by mouth.
  Irinotecan is approved for adult subjects with some forms of colorectal cancer. It is also considered "investigational" for brain tumors. Irinotecan dose will depend on your height & weight. Irinotecan will be given intravenously over 90 min on days 1, 14 & 28 of 6wk cycle.
  You will be seen in clinic approximately every 42 days for 1st 3 cycles of study drug, & then every other cycle thereafter. Your brain MRI examination will be done within 1 wk prior to completion of cycles 1-3, & then within 1 week prior to completion of every other cycle.
  Other Names: SU011248-Sutent-Sunitinib; Irinotecan-CPT 11-Camptosar

SUMMARY:
Primary Objectives To determine maxi tolerated dose & dose limiting toxicity of SU011248 + Irinotecan in recurrent MG pts not on EIAEDs To characterize safety & tolerability of SU011248 + Irinotecan among pts w recurrent MG Secondary Objectives To evaluate pharmacokinetic profile of SU011248 & Irinotecan when co-administered in pts w MG To evaluate anti-tumor activity of SU011248 + Irinotecan

DETAILED DESCRIPTION:
Primary interest for combining SU011248 w irinotecan in malignant glioma pts derives from dramatic anti-tumor activity recently demonstrated among RMG pts treated w humanized anti-VEGF monoclonal antibody, bevacizumab, when combined w irinotecan. 63 percent radiographic response rate was observed following treatment w regimen every other wk, & median progression-free survival was 23wks. Similar enhancement of chemo activity by VEGF-directed therapy w bev has been previously demonstrated for colorectal & lung cancer pts. SU011248 is being evaluated in current regimen because it may exert more potent anti-angiogenic effect than bev among MG pts due to its ability to inhibit PDGFR-mediated pericyte stabilization in tumor neovasculature.

Current proposed ph I study is designed to determine MTD & DLT of SU011248 when combo w irinotecan for pts w RMG. Both SU01148 & irinotecan are known to be metabolized by CYP3A4 cytochrome system. Current study will limit enrollment to pts who are not on CYP3A4-enzyme inducing anti-epileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Pts confirmed GBM, GS, AA, AO & AOA w recurrent disease following standard therapy consisting of at least external beam XRT & temo chemo
* Pts not had tumor biopsy <1 week/surgical resection <2 weeks prior to starting study drug
* Pts should be on non-increasing dose of steroids >7 days prior to obtaining baseline Gd-MRI of brain
* Age >18yrs
* KPS >70
* ANC >1.5 x 10 9/L
* Hgb >9 g/dL
* Platelets >100 x 10 9/L
* AST/SGOT & ALT/SGPT <2.5 x ULN
* Serum bilirubin <1.5 x ULN
* Serum CA <12 mg/dL
* Serum creatinine <1.5 x ULN/measured 24-hr CrCl>50mL/min/1.73m^2
* Pt has ability to understand & provide signed informed consent that fulfills IRB guidelines

Exclusion Criteria:

* Prior gr3/>toxicity/failure to CPT-11 therapy
* Prior Sunitinib malate therapy
* Concurrent administration of EIAEDs
* Major surgery <2 weeks of enrollment
* History of impaired cardiac function
* Other clinically significant cardiac diseases
* Uncontrolled diabetes
* Active/uncontrolled infection requiring intravenous antibiotics
* Impairment of GI function/GI disease that may significantly alter absorption of Sunitinib malate Sutent
* Acute/chronic liver/renal disease
* Cerebrovascular accident/transient ischemic attack <6mths of study enrollment
* Pulmonary embolism <6mths of study enrollment
* Pre-existing thyroid abnormality w thyroid function that can not be maintained in normal range w medication
* Pts taking warfarin sodium
* Pts have received chemo ≤4wks to starting study drug unless they have fully recovered from all anticipated side effects of such therapy
* Pts have received immunotherapy ≤2wks to starting study drug/have not recovered from side effects of such therapy
* Pts have received investigational drugs ≤2wks to starting study drug unless they have fully recovered from all anticipated side effects of such therapy
* Pts have received XRT ≤4wks to starting study drug unless they have fully recovered from all anticipated side effects of such therapy
* Pts have undergone major non-CNS surgery ≤2wks to starting study drug/pts who have not recovered from side effects of such therapy
* Cardiac pacemaker
* Ferromagnetic metal implants other than those approved as safe for use in MR scanners
* Claustrophobia
* Obesity
* Female pts who are pregnant/breast feeding/adults of reproductive potential not employing effective method of birth control
* Known diagnosis of HIV
* History of another primary malignancy that is currently clinically significant/currently requiring active intervention
* Pts unwilling to/unable to comply w protocol
* Existing intra-tumoral hemorrhage
* Concurrent participation in another clinical trial except for supportive care/non-treatment trials
* Other severe acute/chronic medical/psychiatric condition/lab abnormality that may increase risk associated w study participation/study drug administration/ may interfere w interpretation of study results, & in judgment of investigator would make subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine MTD & DLT of SU011248 + Irinotecan in pts w RMG not on EIAEDs | 6 months

SECONDARY OUTCOMES:
Demographic & baseline characteristics | 6 months
Efficacy observations & measurements | 6 months
Safety observations & measurements | 6 months
PK measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/